CLINICAL TRIAL: NCT05120713
Title: The Influence of Noradrenergic Activity on Attentional Control in Younger and Older Adults
Brief Title: Noradrenergic Activity and Attention
Acronym: NAA
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Mara Mather, Principal Investigator, University of Southern California
Other Study IDs: UP-21-00711
Record Dates: First submitted 2021-10-13; First posted 2021-11-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: attention; arousal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young Adults: Young Adults aged 18-35
- Older Adults: Older Adults aged 50-80

SUMMARY:
Older adults demonstrate increased distractibility by task-irrelevant information which contributes to general cognitive impairment. However, it is yet unclear how changes in noradrenergic activity during aging influences attentional control. In the current study, tonic noradrenergic activity will be increased or decreased to investigate its behavioral and neural effects on attentional control.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Aged between 18-35 or 50-80
* Have normal or corrected-to-normal vision and hearing, and normal color vision
* Have a mobile phone and email address

Exclusion Criteria:

* Non-English speakers
* Currently practicing any relaxation, meditation, or breathing technique for more than an hour per week
* Have participated in studies measuring attentional capture in the past year
* Experiencing symptoms of dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young adults will be recruited from the student population at the University of Southern California. Older adults will be recruited from a volunteer registry.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USC Leonard Davis School of Gerontology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, data in de-identified form will be shared using the Open Science Framework and/or OpenNeuro Databases which are free and open platforms for sharing and archiving scientific data.
Time Frame: Data will be made available at the end of the experiment, indefinitely.
Access Criteria: Data will be uploaded to scientific data archiving platforms.

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Adults: Young Adults aged 18-30
Period: Overall Study
Arm/Group | Young Adults | Older Adults
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Adults | Older Adults | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Customized [Count of Participants; unit: Participants]
  Age: 18 to 30 years old inclusive | 70 | 0 | 70
  Age: 50 to 80 years old inclusive | 0 | 70 | 70
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 21 | 20 | 41
  Sex: Female | 48 | 50 | 98
  Sex: Choose not to report | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 10 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 15 | 47 | 62
  More than one race | 10 | 4 | 14
  Unknown or Not Reported | 10 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Initial Eye-movements Toward Target and Distractor Shapes Measured by an Eye-tracker
Description: The oculomotor suppression effect is a lower likelihood that salient display items will be the target of the initial eye movement in a visual search task compared to nonsalient display items. This effect is calculated from the percentage of first saccades toward a non-target stimuli subtracted by the percentage of first saccades toward the distractor stimuli. Greater % of first saccades toward the target would demonstrate better goal-directed attentional control and greater % of first saccades toward the distractor would demonstrate increased distractibility. Thus, a greater oculomotor suppression effect would demonstrate an increased ability to inhibit salient information that is irrelevant to the task.
Time Frame: Calculated once at the end of the 1 day experiment
Population: Both young and older adults completed the experiment at baseline and under increased arousal (order counterbalanced).
Measure: Mean (Standard Error); unit: percentage of first saccades
Groups:
- Young Adults Baseline: Young adults aged 18-30 under no intervention
- Older Adults Basline: Older adults aged 50-80 under no intervention
- Young Adults + Arousal: Young adults aged 18-30 years older during the threat of shock block
- Older Adults + Arousal: Older adults aged 50-80 years older during the threat of shock block
Arm/Group | Young Adults Baseline | Older Adults Basline | Young Adults + Arousal | Older Adults + Arousal
Number analyzed (Participants) | 70 | 70 | 70 | 70
percentage of first saccades | 3.8 (0.3) | 4.4 (1.2) | 3.6 (0.7) | 4.5 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for one day during when the subject came into the lab to complete the experiment.
Description: The intervention has minimal risk and expect no serious adverse events or mortality.
Arm/Group | Young Adults | Older Adults
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT05120713/Prot_SAP_000.pdf